CLINICAL TRIAL: NCT01183143
Title: A Multicentre, Open-label, Non-comparative Phase IIIb Study to Evaluate the Acceptability of GONAL-f® Prefilled Liquid Formulation Administered by Pen in an Outpatient Setting for Ovarian Stimulation
Brief Title: Convenience and Safety of Assisted Reproductive Technology Procedures Using a Gonal-F Filled by Mass (Fbm) Liquid Formulation Applied by Pen for Ovulation Induction and In-vitro Fertilization
Acronym: Prestyje
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMP 25040
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Infertility; Ovulation Induction; In-Vitro Fertilization
Keywords: Infertility; Ovulation induction; Gonal-F; Follitropin alpha; Controlled ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Glycoprotein Hormones, alpha Subunit

ARMS (1):
- GONAL-f® (Experimental)
  Interventions: Drug: GONAL-f®

INTERVENTIONS:
Drug: GONAL-f® — GONAL-f® will be administered subcutaneously to subjects between Day 2 and Day 5 of their cycle with a starting dose of 75 International Units (IU) per day for subjects who undergo ovulation induction (OI)/artificial insemination (IUI) and between 150 and 225 IU per day for subjects who undergo in-vitro fertilization (IVF). For subjects who undergo OI/IUI, the dose will be increased by 37.5 IU after Day 14 up to Week 4 if no ovarian response is observed.
  Other Names: Follitropin alpha

SUMMARY:
This was a prospective, open-label, non-comparative, Phase IIIb trial to assess the convenience, safety and efficacy of the new Gonal-F fbm [recombinant follicle stimulating hormone (r-FSH)] liquid formulation, in common setting for ovulation induction (OI) and also in in-vitro fertilization (IVF).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged between 18 and 43 years
* Ambulatory subjects
* Subjects who are willing to get pregnant and are infertile, that justifies ovarian stimulation treatment for mono-/pauci-follicular development (OI or IUI) or multiple follicular development for IVF/Intracytoplasmic Sperm Injection (ICSI) procedures
* Subjects who are able to communicate well with the investigator and to comply with the requirements of the entire study
* Subjects who have given written informed consent, prior to treatment

Exclusion Criteria:

* Subjects with enlarged ovaries or cysts unrelated to polycystic ovaries
* Subjects with extra-uterine pregnancy during the last 3 months
* Subjects with several endometriosis (Grade III & IV)
* Subjects with history of severe ovarian hyperstimulation syndrome
* Subjects with history of thromboembolic event
* Subjects with malformative uterine pathology that could disturb either implantation or pregnancy processes
* Subjects with premature menopause
* Subjects with gynecological bleeding of unknown origin
* Subjects with ovarian, uterine, or mammary cancer
* Subjects with tumors of the hypothalamus or the pituitary glands
* Subjects with history of serious allergy or atopic asthma disease
* Subjects with known allergic reaction against one of the Follicle Stimulating Hormone (FSH) and ingredients,
* Ongoing pregnant, or breast feeding subjects
* Subjects who have participated in a trial during the last 3 months

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 2004-05-11 (Actual); Primary Completion 2006-03-02 (Actual); Study Completion 2006-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please Contact the Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- GONAL-f®: GONAL-f® was administered subcutaneously to subjects between Day 2 and Day 5 of their cycle with a starting dose of 75 International Units (IU) per day for subjects who underwent ovulation induction (OI)/ artificial insemination (IUI) and between 150 and 225 IU per day for subjects who underwent in-vitro fertilization (IVF). For subjects who underwent OI/ IUI the dose was increased by 37.5 IU after Day 14 up to Week 4 if no ovarian response was observed.
Period: Overall Study
Arm/Group | GONAL-f®
Started | 215
Intention to Treat (ITT) Population | 204 (ITT=Subjects who received at least 1 dose of the investigational medicinal product (IMP).)
Completed | 65
Not Completed | 150
Not completed — Protocol Violation | 115
Not completed — Withdrawal by Subject | 19
Not completed — Subject Questionnaires not returned | 5
Not completed — Subjects enrolled, but not treated | 11

BASELINE CHARACTERISTICS:
Population: The ITT population included all the subjects who received at least 1 dose of the IMP.
Arm/Group | GONAL-f®
Number analyzed (Participants) | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Self-administered the Investigational Medicinal Product (IMP)
Description: Number of subjects who self-administered the IMP were presented in this outcome measure.
Time Frame: Up to 1 year
Population: The ITT population included all the subjects who received at least 1 dose of the IMP.
Measure: Number; unit: subjects
Arm/Group | GONAL-f®
Number analyzed (Participants) | 204
subjects | 159

2. Secondary Outcome: Global Evaluation of the GONAL-f® Prefilled Pen by the Investigator
Description: Investigator evaluated the use of GONAL-f® prefilled pen in subjects as very satisfactory, satisfactory and average satisfaction.
Time Frame: Up to 1 year
Population: The ITT population included all the subjects who received at least 1 dose of the IMP. Here "Overall Number of Subjects Analyzed" signifies those subjects who were evaluable for this outcome.
Measure: Number; unit: subjects
Arm/Group | GONAL-f®
Number analyzed (Participants) | 195
subjects
  Very satisfactory | 101
  Satisfactory | 93
  Average satisfaction | 1

3. Secondary Outcome: Evaluation of the Information Given to the Subjects on the Pen's Utilization
Description: Subjects were provided with the information on Pen's utilization via training session and in the form of information brochure. Subjects assessed both the methods using the following responses: satisfactory, satisfactory, unsatisfactory and very unsatisfactory.
Time Frame: Up to 1 year
Population: The ITT population. Here "Overall Number of Subjects Analyzed" signifies those subjects who were evaluable for this outcome and "Number Analyzed" signifies those who were evaluable for the specified category.
Measure: Number; unit: subjects
Arm/Group | GONAL-f®
Number analyzed (Participants) | 195
subjects
  Training Session: Very satisfactory: number analyzed (Participants) | 190
  Training Session: Very satisfactory | 89
  Training Session: Satisfactory: number analyzed (Participants) | 190
  Training Session: Satisfactory | 95
  Training Session: Unsatisfactory: number analyzed (Participants) | 190
  Training Session: Unsatisfactory | 5
  Training Session: Very unsatisfactory: number analyzed (Participants) | 190
  Training Session: Very unsatisfactory | 1
  Information brochure: Very satisfactory | 95
  Information brochure: Satisfactory | 89
  Information brochure: Unsatisfactory | 9
  Information brochure: Very unsatisfactory | 2

4. Secondary Outcome: Duration of Ovarian Stimulation With GONAL-f®
Description: Stimulation duration was defined as the duration (in days) for which subjects underwent GONAL-f® treatment.
Time Frame: Up to 1 year
Population: The ITT population included all the subjects who received, at least 1 dose of the IMP.
Measure: Median (Full Range); unit: days
Arm/Group | GONAL-f®
Number analyzed (Participants) | 204
days | 10 [3 to 26]

5. Secondary Outcome: Mean Number of Embryos Transferred
Time Frame: End of Stimulation period (up to a maximum 26 days)
Population: The ITT population included all the subjects who received at least 1 dose of the IMP. Here "Number of Participants Analyzed" signifies those subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | GONAL-f®
Number analyzed (Participants) | 119
embryos | 1.8 (0.7)

6. Secondary Outcome: Total and Average Daily Dose of GONAL-f®
Time Frame: Up to 26 days
Population: The ITT population included all the subjects who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: International Units (IU)
Arm/Group | GONAL-f®
Number analyzed (Participants) | 204
International Units (IU)
  Total dose | 1527 (964)
  Daily dose | 149.5 (75.9)

7. Secondary Outcome: Pregnancy Rate in Subjects Receiving Stimulation by Ovulation Induction (OI) or Artificial Insemination (IUI)
Description: Pregnancy rate was defined as the percentage of subjects with diagnosis of pregnancy, who underwent OI/IUI. Clinical pregnancy: Evidence of pregnancy by clinical or ultrasound parameters at 12 weeks after fertilization. Biochemical pregnancy: Evidence of conception based only on biochemical data in the serum or urine before ultrasound evidence of a gestational sac. Ongoing pregnancy was defined when the pregnancy had completed 20 weeks of gestation.
Time Frame: Up to 20 Weeks of Gestation
Population: The ITT population included all the subjects who received, at least 1 dose of the IMP. "Number of Participants Analyzed" signifies ITT (OI/IUI) subjects who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GONAL-f®
Number analyzed (Participants) | 85
Percentage of subjects
  Clinical pregnancy | 16.5 [8.6 to 24.4]
  Biochemical pregnancy | 16.5 [8.6 to 24.4]
  Ongoing pregnancy | 16.5 [8.6 to 24.4]

8. Secondary Outcome: Number of Subjects With Live Birth
Description: Number of subjects whose stimulation with the IMP resulted in the birth of a baby were reported.
Time Frame: End of Gestation period, assessed up to a maximum of 1 year
Population: Per Protocol (PP) population was defined as the group of subjects who completed the study, having returned their completed questionnaire and who did not present any major protocol deviations.
Measure: Number; unit: subjects
Arm/Group | GONAL-f®
Number analyzed (Participants) | 181
subjects | 41

9. Secondary Outcome: Number of Subjects With Local Tolerance at GONAL-f ® Injection Site as Assessed by Investigator
Description: Local tolerance at the GONAL-f ® injection site was assessed for the presence of pain, swelling/welt, redness, itch and haematoma.
Time Frame: Up to 1 year
Population: ITT population included all the subjects who received at least 1 dose of the investigational medicinal product.
Measure: Number; unit: subjects
Arm/Group | GONAL-f®
Number analyzed (Participants) | 204
subjects
  Pain | 32
  Swelling/welt | 3
  Redness | 34
  Itch | 8
  Haematoma | 41

10. Secondary Outcome: Number of Subjects With at Least 1 Adverse Event
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerged or worsened relative to baseline (i.e. present at the initial study visit) during a clinical study with an investigational product, regardless of causal relationship and even if no investigational product has been administered.
Time Frame: Up to 1 year
Population: The tolerance analysis set included of all the subjects who were presented at the inclusion visit.
Measure: Number; unit: subjects
Arm/Group | GONAL-f®
Number analyzed (Participants) | 215
subjects | 36

11. Secondary Outcome: Number of Subjects Taking at Least 1 Concomitant Treatment
Time Frame: Up to 1 year
Population: The tolerance analysis set included of all the subjects who were presented at the inclusion visit.
Measure: Number; unit: subjects
Arm/Group | GONAL-f®
Number analyzed (Participants) | 215
subjects | 28

ADVERSE EVENTS:
Description: As per the planned analysis, data was collected for the tolerance population (overall population) irrespective of the type of stimulation. The tolerance population consisted of all the subjects who were presented at the inclusion visit.
Arm/Group | GONAL-f®
Serious Adverse Events (participants affected / at risk) | 6/215
Other Adverse Events (participants affected / at risk) | 36/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GONAL-f® (N=215)
Abortion spontaneous NOS (Pregnancy, puerperium and perinatal conditions) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2
Placental, amniotic and cavity disorders (Pregnancy, puerperium and perinatal conditions) | 1
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GONAL-f® (N=215)
Abdominal pain upper (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Injection site erythema (General disorders) | 4
Injection site haemorrhage (General disorders) | 15
Injection site pain (General disorders) | 4
Injection site pruritus (General disorders) | 2
Pelvic infection (Infections and infestations) | 1
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Abortion spontaneous NOS (Pregnancy, puerperium and perinatal conditions) | 3
Metrorrhagia (Reproductive system and breast disorders) | 1
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 4
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhoids (Vascular disorders) | 1
Venous insufficiency (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other